CLINICAL TRIAL: NCT01098422
Title: A Phase II Study of Yttrium-90 Radioactive Resin Microspheres in the Treatment of Colorectal Adenocarcinoma Metastatic to the Liver After Failure of First-Line Combination Chemotherapy
Brief Title: A Study of Yttrium-90 Radioactive Resin Microspheres to Treat Colorectal Adenocarcinoma Metastatic to the Liver
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Halted due to slow enrollment
Sponsor: Tony Reid, M.D., Ph.D. (Other)
Collaborators: Sirtex Medical (Industry)
Responsible Party: Sponsor-Investigator, Tony Reid, M.D., Ph.D., Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 071960
Record Dates: First submitted 2010-04-01; First posted 2010-04-02 (Estimated); Results first posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Colorectal Neoplasms; Liver Neoplasms
Keywords: liver; colorectal; metastasis; carcinoma; Yttrium-90; microspheres
MeSH Terms: conditions — Colorectal Neoplasms; Liver Neoplasms; Neoplasm Metastasis; Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Yttrium-90 Radioactive Resin Microspheres (Experimental): Yttrium-90 Radioactive Resin Microspheres
  Interventions: Device: Yttrium-90 Radioactive Resin Microspheres

INTERVENTIONS:
Device: Yttrium-90 Radioactive Resin Microspheres — An injectable formulation of the radioisotope yttrium-90 encapsulated in resin microspheres with potential antineoplastic activity.

SUMMARY:
The purpose of this study is to determine the effectiveness of radioactive microsphere infusion as a treatment for liver metastases from colon or rectal cancer. The investigators hypothesis is that the administration of microspheres between first and second line chemotherapy will increase progression-free survival time by about 2.5 months and may also improve tumor response rates to subsequent second line chemotherapy.

DETAILED DESCRIPTION:
This is a phase II, single-arm study of Yttrium-90 (Y-90) radioactive resin microspheres in the treatment of colorectal adenocarcinoma metastatic to the liver in patients who have had progressive disease through first line combination chemotherapy or have otherwise failed first line chemotherapy due to toxicity. Expected enrollment at University of California, San Diego (UCSD) is approximately 34 subjects.

The dose of Yttrium-90 radioactive resin microspheres is calculated based on body surface area (to estimate normal liver volume), percentage of total liver represented by the targeted lobe, and percentage of the lobe that is occupied by tumor, corrected for percentage lung shunt. The prescribed dose, calculated by the nuclear medicine physician, will be delivered by the interventional radiologist using the standard delivery system with frequent fluoroscopic monitoring to assure ante grade blood flow immediately after treatment. Additional current standard practice includes obtaining a nuclear medicine scan of the patient immediately after each therapeutic Yttrium-90 microspheres administration to prove delivery of the agent to the targeted portion of the liver and absence of either extra-hepatic Yttrium-90 delivery or free Yttrium-90.

Blood samples will be obtained one week after the first treatment with microspheres. If the patient has bi-lobar disease and the results of lab tests meet protocol specified criteria, the dose will be repeated in the initially-untreated lobe. If the lab tests do not meet protocol specified criteria (i.e. study inclusion/exclusion criteria), the treatment will be deferred for fourteen days and labs repeated. If they are then within parameters, the patient will receive the second dose. If they are not within parameters, the patient will proceed to chemotherapy.

Patients will remain off chemotherapy after their final microspheres treatment for a minimum of three weeks. Second line treatment options include FDA approved anti-neoplastic agents used in colorectal cancer metastatic to the liver with the exception of bevacizumab and capecitabine, which has been less rigorously studied with relation to Yttrium-90 radioactive microspheres and therefore will not be used. When patients are found to have progressive disease while receiving second line chemotherapy, they will then undergo a comprehensive clinical, laboratory, and imaging assessment and enter the follow-up phase in which they are assessed every five to seven months until death or withdrawal of consent.

A contrast enhanced ultrasound (CEUS) will be performed pre microsphere treatment (within 14 days), post microsphere treatment (2 weeks, 4 weeks, 8 weeks and 12 weeks post the microsphere treatment). If patients require two treatments with microspheres, they will be evaluated 2, 4, 8 and 12 weeks post the second treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed colorectal carcinoma. Liver metastasis will be confirmed by either PET scan or biopsy.
* Ability to understand and willingness to sign written informed consent
* Minimum of 18 years of age
* Liver dominant metastases measurable by CT or MRI and therefore amenable to serial assessment using RECIST criteria
* Progressive disease of metastatic colorectal carcinoma on first line combination chemotherapy with a 5-fluorouracil/leucovorin with oxaliplatin (FOLFOX) based regimen (Folinic Acid, Oxaliplatin and Fluorouracil)or failure of first line chemotherapy due to toxicity
* Candidate for second line chemotherapy with a fluorouracil, leucovorin, and irinotecan (FOLFIRI) regimen. Per standard of care, second line chemotherapy will not include Bevacizumab.
* Karnofsky Performance Score (KPS) of 70% or greater
* Life expectancy of greater than or equal to four months by investigator estimation
* Females with negative urine or serum pregnancy test
* Effective double barrier contraception for a minimum of two months following the final infusion of microspheres
* Patients who are not candidates for transarterial chemoembolization (TACE), thermal ablation or surgical resection

Exclusion Criteria:

* Dominant extra-hepatic disease including cerebral metastases or other extra-hepatic metastases that are symptomatic
* Large volume ascites assessed by cross sectional CT imaging
* Any chemotherapy < 4 weeks prior to the first microsphere treatment
* Anticipated to need Avastin chemotherapy within eight weeks of day M1
* Absolute neutrophil count (ANC) < 1.5 x 109/L
* Platelets (PLT) < 60,000/mm3
* Hemoglobin (Hgb) < 9.0 gm/dL
* Prothrombin time (PT) or Partial Prothrombin time (PTT) > upper limit of normal (ULN)
* Serum Creatinine > 2.0 mg/dL
* Forced expiratory volume (FEV1) < 1L by baseline pulmonary function tests (ordered if investigator judges it to be clinically indicated)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 5 times upper limits of normal (ULN) or total bilirubin > 2.0 mg/dL
* History of incompetent sphincter of oddi (e.g.: sphincterotomy, biliary-enteric anastamosis, or percutaneous biliary drain)
* Severe hypoalbuminemia (albumin < 2.0 g/dL)
* Alkaline phosphatase > 2.5 times ULN
* Greater than 20% lung shunting (determined by the MAA - Tc 99 nuclear medicine lung shunt scan)
* Pre assessment angiogram and MAA scan demonstrating any uncorrectable activity in the stomach, bowel or pancreas
* Major surgery < 4 weeks prior to the first microsphere treatment
* Female who is pregnant or nursing
* Men and women of childbearing potential wishing to conceive < 2 months following the completion of the microsphere portion of the study.
* Any investigational agent administered < 4 weeks prior to microsphere treatment
* A known history of hepatitis B or hepatitis C
* Known hypersensitivity to any component of microsphere infusion
* History of, or current coagulation or bleeding disorder
* History of significant hepatic cirrhosis, fibrosis or hemochromatosis
* History of malignancy, other than colorectal cancer, within five years of the start of study participation, except in situ cervical or skin cancer
* Active severe infection or any other concurrent disease or medical conditions that are likely to interfere with the study as judged by the investigator
* Prior treatment with radioactive microspheres or external beam radiation therapy to the liver
* Prophylactic anticoagulation and nonsteroidal antiplatelet drugs are only a contraindication, if the PT/PTT are above the ULN. Plavix (clopidogrel) will need to be stopped 5 days prior to the hepatic-angiogram and the microsphere procedures, then started the next day.
* History of right to left, bi-directional or transient right to left cardiac shunts, worsening or clinically unstable congestive heart failure, acute myocardial infarction or acute coronary syndromes serious ventricular arrhythmias or high risk for arrhythmias due to prolongation of the QT interval, respiratory failure as manifested by signs or symptoms of carbon dioxide retention or hypoxemia or severe emphysema, pulmonary emboli or other conditions that causes pulmonary hypertension due to compromised pulmonary arterial vasculature

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tony Reid, MD, PhD, Principal Investigator — University of California, San Diego
Locations (2):
- United States (2):
  - The Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - UCSD Medical Center, San Diego, California

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Yttrium-90 Radioactive Resin Microspheres
Started | 10
Completed | 9
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Yttrium-90 Radioactive Resin Microspheres
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 5
Age, Continuous [Mean (Full Range); unit: years] | 64.3 [52 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — United States California
  Participants
    United States | 10

OUTCOME MEASURES:

1. Primary Outcome: PFS
Description: Progression-free survival assessed by Response Evaluation Criteria in Solid Tumors (RECIST) criteria using Computerized Tomography (CT) assessment of tumor(s)
Time Frame: 2 years
Measure: Median (Standard Deviation); unit: Months
Arm/Group | Yttrium-90 Radioactive Resin Microspheres
Number analyzed (Participants) | 9
Months | 7.6 (12.7)

2. Secondary Outcome: Percentage of Participants Achieving Overall Survival at 6 Months
Description: Overall survival assessed at 6 months since diagnosis of progression on first-line therapy
Time Frame: 6 Months
Measure: Number; unit: percent
Arm/Group | Yttrium-90 Radioactive Resin Microspheres
Number analyzed (Participants) | 9
percent | 78

3. Secondary Outcome: Number of Participants With Responses as Determined by RECIST Criteria Using CT or Magnetic Resonance Imaging (MRI) Assessment
Description: Tumor response rate as determined by RECIST criteria using CT or Magnetic Resonance Imaging (MRI) assessment of tumor size every 3 months
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Yttrium-90 Radioactive Resin Microspheres
Number analyzed (Participants) | 9
participants | 9

4. Secondary Outcome: Adverse Events
Description: Number of adverse events by grade
Time Frame: 1 years
Measure: Number; unit: Events
Arm/Group | Yttrium-90 Radioactive Resin Microspheres
Number analyzed (Participants) | 9
Events
  Nausea | 10
  Emesis | 7
  Pain | 13
  Weight Loss | 4
  Fatigue | 39
  Fever | 2
  Bilirubin | 4
  Alk Phos | 20.5
  ALT | 1
  AST | 1

5. Secondary Outcome: 60 Day All-cause Mortality Rate
Description: Number of Participants with 60 Day All-cause Mortality
Time Frame: 60 days
Measure: Number; unit: participants
Arm/Group | Yttrium-90 Radioactive Resin Microspheres
Number analyzed (Participants) | 9
participants | 0

ADVERSE EVENTS:
Arm/Group | Yttrium-90 Radioactive Resin Microspheres
All-Cause Mortality (participants affected / at risk) | 9/9
Serious Adverse Events (participants affected / at risk) | 9/9
Other Adverse Events (participants affected / at risk) | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Yttrium-90 Radioactive Resin Microspheres (N=9)
Nausea (Gastrointestinal disorders) | 1 (1)
Emesis (Gastrointestinal disorders) | 1 (1)
Fatigue (Gastrointestinal disorders) | 4 (4)
Alk Phos (Hepatobiliary disorders) | 2 (2)
Bilirubin (Hepatobiliary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes